CLINICAL TRIAL: NCT01820897
Title: Fosfomycin-Trometamol in Urinary Tract Infection Prophylaxis After Kidney Transplantation. Randomized Controlled Trial.
Brief Title: Efficacy of Fosfomycin-Trometamol in Urinary Tract Infection Prophylaxis After Kidney Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JOSE MANUEL ARREOLA GUERRA (Other)
Collaborators: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor-Investigator, JOSE MANUEL ARREOLA GUERRA, Nephrologist and Internal medicine physician, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Organization: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UTIPROPH-625
Record Dates: First submitted 2013-03-26; First posted 2013-03-29 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Urinary Tract Infection; Asymptomatic Bacteriuria; Allograft Rejection; Microbiologic Resistance; Hospitalization
MeSH Terms: conditions — Urinary Tract Infections | interventions — Fosfomycin; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fosfomycin-Trometamol, Sulfamethoxazole trimethoprim, placebo (Experimental): Fosfomycin-Trometamol 3 grams every 10 days for 6 months Plus Sulfamethoxazole trimethoprim 800/160 mg monday, wednesday and friday for 6 months Plus Placebo of Sulfamethoxazole trimethoprim Tuesday,thursday, saturday and sunday for 6 months.
  Interventions: Drug: Fosfomycin-Trometamol
- Sulfamethoxazole trimethoprim, placebo (Active Comparator): Sulfamethoxazole trimethoprim 800/160 mg every day for 6 months plus Placebo of Fosfomicyn-trometamol every 10 days for 6 months
  Interventions: Drug: Sulfamethoxazole trimethoprim

INTERVENTIONS:
Drug: Fosfomycin-Trometamol
  Arms: Fosfomycin-Trometamol, Sulfamethoxazole trimethoprim, placebo
Drug: Sulfamethoxazole trimethoprim
  Arms: Sulfamethoxazole trimethoprim, placebo

SUMMARY:
Urinary tract infections (UTI) are the most common complications after kidney transplantation. Most series have reported incidence between 20 to 50% during the first year. In the most recent report from our center the incidence was 36.6% during the first 6 months after transplantation.

The clinical consequence in the graft survival and the association with immunological rejection has not been well defined. Nevertheless, the association of UTI with high rate of hospitalization and their costs are widely recognized. There is paucity of trials, specially randomized and controlled, comparing antibiotic prophylaxis in this group of patients. In a recently published metaanalysis Green et al. (Transpl Infect Dis. 2011 Oct;13(5):441-7) found only 6 clinical trials well designed, the conclusion was that antibiotic prophylaxis reduced the incidence of UTI and the risk of sepsis. Based in this information, the KDIGO guidelines in transplantation recommend the prophylaxis for UTI with sulfamethoxazole-trimethoprim (SMT). Nevertheless, the rate of bacterial resistance to SMT has been reported above 50% in almost all the series.

Fosfomycin-trometamol (FT) is a wall antibiotic (piruvil-tranferase inhibitor) that has shown a good bioavailability, especially in the urinary tract. It has shown a wide antibacterial spectrum, but the important target seems to be enteric bacilli particularly Escherichia coli (the most prevalent cause of UTI). FT has also shown a very good activity against E. coli producer of Extended Spectrum Betalactamases. Recently, the rate of these multi-drug resistant bacteria has increased in our center as evidence of worldwide distribution. In addition, the rate of FT resistance has been stable during the last years (<3%). This phenomenon could be explained because of the properties of this antibiotic, the most important one seems to be related with the unique mechanism of action and the lack to propagate the mechanisms of resistance at least in E. coli. There is only one clinical trial (randomized and controlled), which compared FT with placebo in UTI prophylaxis; 317 women with recurrent UTI (three by year) were included. They found rates of 0.14 and 2.9 episodes/patient/year, respectively (p<0.001). Furthermore, there was no FT resistance during the follow up.

Our hypothesis is that in the first six months after kidney transplantation, UTI prophylaxis with FT will show greater efficacy in comparison with SMT. Considering the incidence of UTI in our center (36.6%) and the rate of UTI in the unique trial of prophylaxis with FT (14%), 65 patients will be needed by group of treatment to demonstrate a difference of 22% in the incidence of UTI, with a power of 80% and confidence level of 95%. The primary outcome is the incidence and rate of UTI during the first six months after kidney transplantation. The secondary outcomes are, the hospitalization rate, antibiotic resistance rate, rejections and titer and number of de novo donor specific antibodies.

The investigators propose a randomized, double blind, placebo controlled trial to compare FT with SMT in the efficacy and safety to prevent UTI during the first six months after kidney transplantation. The investigators will include patients from two tertiary-care transplant centers. Recruiting and the randomization will be carried out separately by center and gender (because female patients have a greater risk of UTI). The medical visits will be scheduled monthly and include general laboratory, urine culture and information gathering about antibiotic side effects as well as adherence. Rejection rate and the number and titers of de novo donor specific antibodies (secondary outcome) will be obtained according to the standard of care of the institutional kidney transplantation follow up. These include kidney biopsy at days 0 and 90 after transplantation, as well as determination of donor specific antibodies after sixth months of follow up. Graft biopsy is also performed whenever graft dysfunction exists in the absence of an identifiable cause (infection, urinary graft obstruction).

ELIGIBILITY:
Inclusion Criteria:

* Patients transplanted in the National Institute of medical Sciences and Nutrition Salvador Zubiran and in the National Institute of Cardiology Ignacio Chavez

Exclusion Criteria:

* Allergy to Fosfomycine-trometamol or Sulfamethoxazole-trimethoprim

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Urinary tract infection incidence in the first six months after kidney transplantation | Six months after kidney transplantetion
  We also will determine the rate of urinary tract infection in the same period. The definition of urinary tract infection include asymptomatic bacteriuria defined by urinary culture with more than 100,000 colonies.

SECONDARY OUTCOMES:
Complications related to the intervention, including rate of microbiological resistance. | Six months after kidney transplantation

OTHER OUTCOMES:
Rate of allograft rejection | Six months after kidney transplantation
Behavior of de novo donor specific antibody (number and titles) | Six months after kidney transplantation
  All the patients in the pre transplant evaluation have determination of donor specific antibody. The behavior of number and titles of these antibodies will be compared with a new measure at the end of followup (six months). Nevertheless if the patient previously has suspected humoral rejection, this determination would be taken in this moment, because is a diagnosis criteria of humoral rejection.

CONTACTS AND LOCATIONS:
Locations (2):
- Mexico (2):
  - National Institute of Medical Sciences and Nutrition Salvador Zubiran, Mexico City, Mexico City
  - National Institute of Medical Science and Nutrition Salvador Zubiran, México, Mexico DF

REFERENCES:
- [Derived] Arreola-Guerra JM, Rosado-Canto R, Alberu J, Maravilla E, Torres-Gonzalez P, Criollo E, Perez M, Mancilla E, Arvizu M, Morales-Buenrostro LE, Vilatoba-Chapa M, Sifuentes-Osornio J. Fosfomycin trometamol in the prophylaxis of post-kidney transplant urinary tract infection: A controlled, randomized clinical trial. Transpl Infect Dis. 2018 Oct;20(5):e12980. doi: 10.1111/tid.12980. Epub 2018 Sep 10. PMID 30133928